CLINICAL TRIAL: NCT00072631
Title: A Phase II, Open-label, Intra-patient Dose-escalation Study of Erlotinib in Patients With Advanced Non-small Cell Lung Cancer Who Have Failed Prior Chemotherapy
Brief Title: Erlotinib (Tarceva (Trademark), OSI-774) in Treating Patients With Advanced Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: OSI Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSI-774-202; Dose to Rash
Record Dates: First submitted 2003-11-05; First posted 2003-11-07 (Estimated); Last update posted 2018-02-08 (Actual); Status verified 2015-06

CONDITIONS: Advanced Non Small Cell Lung Cancer; Failed Prior Chemotherapy
Keywords: Tarceva; erlotinib; NSCLC; Non-Small Cell Lung Cancer; EGFR; OSI-774
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Erlotinib Hydrochloride; Patents as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 erlotinib (Experimental)
  Interventions: Drug: Tarceva (Trademark) (erlotinib HCl, OSI-774)

INTERVENTIONS:
Drug: Tarceva (Trademark) (erlotinib HCl, OSI-774) — Intrapatient dose escalation of oral single agent daily erlotinib until intolerable rash

SUMMARY:
The purpose of this study is to determine if erlotinib will improve disease at doses that produce its characteristic rash in patients with advanced Non-Small Cell Lung Cancer.

DETAILED DESCRIPTION:
Only patients with 0 to 1 performance status on the ECOG scale are eligible.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of Stage IIIB or IV non-small cell lung cancer (histological or cytological).
* Received prior chemotherapy treatment for advanced, metastatic non-small cell lung cancer.
* Measurable disease per RECIST criteria.
* Adequate bone marrow, hepatic and renal function.

Exclusion Criteria:

* Breast cancer or skin cancer at any time in the past or any other cancer in the past 5 years.
* Brain metastases that are unstable, require steroids, are life-threatening or required radiation in the last 28 days.
* Known hypersensitivity to minocycline.
* History of serious cardiac disease that is not controlled.
* Serious eye conditions.
* Prior treatment with inhibitors of EGFR of any kind.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2003-11-05 (Actual); Primary Completion 2007-03-14 (Actual); Study Completion 2007-03-14 (Actual)

PRIMARY OUTCOMES:
Feasibility of intrapatient dose escalation of erlotinib HCI to introduce a characteristic, target rash, and evaluate the effect on objective response rate | 3 years

SECONDARY OUTCOMES:
Feasibility of correlating objective response rate and duration of response to grade of rash | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Institute for Drug Development Cancer Therapy and Research Center, San Antonio, Texas, United States

REFERENCES:
- See also: Link to results on Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/study.aspx?ID=56